CLINICAL TRIAL: NCT03712306
Title: The (Cost) Effectiveness of Increasing Daily Protein Intake to 1.2 Gram Per Kilo Body Weight on Physical Functioning in Community-dwelling Older Adults With a Habitual Daily Protein Intake < 1.0 Gram Per Kilo Body Weight
Brief Title: The (Cost)Effectiveness of Increasing Protein Intake on Physical Funtioning in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: University of Helsinki (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Ilse Reinders, Principal investigator, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 678732
Record Dates: First submitted 2018-07-02; First posted 2018-10-19 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Protein-Energy Malnutrition; Physical Disability
MeSH Terms: conditions — Protein-Energy Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Participants will be randomized intro one of the three study groups.
  Stratification by gender and habitual protein intake (low protein (>=0.9 g/kg aBW/day - <1.0 g/kg aBW/day), very low protein (<0.9 g/kg aBW/day)), since we expect a different intervention effect for participants with a very low baseline habitual protein intake (< 0.9 g/kg aBW/d) compared to participants with a low baseline habitual protein intake (≥ 0.9 g/kg aBW/d), and because of potential differences in how women and men respond to the intervention.
  In case couples participate, we will make sure they will be allocated to the same intervention group. This will ensure no interference between intervention groups. We will randomly select whether the randomization for the intervention group is based on the men or the women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): No intervention. Participants will only receive a brochure on general healthy eating habits.
- Dietary advice (Experimental): Personalized nutritional advice from a registered dietician or nutritionist aimed at increasing protein intake to at least 1.2 g/kg adjusted body weight/d, through intake of regular protein rich food products and provided protein-enriched food products.
  Interventions: Other: Dietary advice
- Dietary advice and advice on timing (Experimental): Personalized nutritional advice from a registered dietician or nutritionist aimed at increasing protein intake to at least 1.2 g/kg adjusted body weight/d, through intake of regular protein rich food products and provided protein-enriched food products, as well as advice regarding the consumption of protein rich food products in close proximity of usual physical activity.
  Interventions: Other: Dietary advice and advice on timing

INTERVENTIONS:
Other: Dietary advice — Dietary advice to increase protein intake to at least 1.2 g/kg adjusted body weight/d
  Arms: Dietary advice
Other: Dietary advice and advice on timing — Dietary advice to increase protein intake to at least 1.2 g/kg adjusted body weight/d plus advice on consuming protein in close proximity of usual physical activity
  Arms: Dietary advice and advice on timing

SUMMARY:
In this RCT with the duration of 6 months among 264 community-dwelling older adults (65+ years) with habitual low protein intake, the investigators will examine the long term (cost) effectiveness of increasing daily protein intake to at least 1.2 gram/kg of adjusted body weight on physical functioning in older adults with low protein intake.

DETAILED DESCRIPTION:
In this RCT with the duration of 6 months the investigators will examine the long term (cost) effectiveness of increasing protein intake to at least 1.2 g/kg adjusted body weight/d on physical functioning in older adults with habitual low protein intake. Additionally, the investigators will examine the combined effect of increasing protein intake to at least 1.2 g/kg adjusted body weight/d and consuming protein in close proximity with regular physical activity on physical functioning in older adults with habitual low protein intake.

Three sub-studies will be conducted, of which the main objectives are to:

1. Examine the effect of persuasive technology on adherence to consumption of protein rich food products in order to increase protein intake to at least 1.2 g/kg adjusted body weight/d, and to the combination of increasing protein intake to at least 1.2 g/kg adjusted body weight/d and consuming protein in close proximity with regular physical activity.
2. Examine the effect of increasing protein intake to at least 1.2 g/kg adjusted body weight/d on faecal and oral microbiota composition in older adults with a habitual low protein intake.
3. Examine the effects of increasing protein intake to at least 1.2 g/kg adjusted body weight/d on food-stimuli related central nervous system satiety and reward responses involved in the regulation of food intake, measured by functional magnetic resonance imaging in older adults with a habitual low protein intake.

   Study design: Randomized controlled trial with the duration of 6 months in two study sites: Amsterdam, the Netherlands and Helsinki, Finland. Stratification by gender and habitual protein intake (low protein (>=0.9 g/kg BW/day - <1.0 g/kg BW/day), very low protein (<0.9 g/kg BW/day)).

   Study population: A total of 264 community-dwelling older adults aged ≥ 65 years with an habitual low protein intake (n=132 at each study site).

   Intervention: This RCT consists of three groups; two intervention groups and one control group. Intervention group 1 (N=44 at each study site) will receive personalized dietary advice aimed at increasing protein intake to at least 1.2 g/kg adjusted body weight/d without changing daily energy intake, by regular foods and by provided protein-enriched food products. Intervention group 2 (N=44 at each study site) receives personalized dietary advice similar to group 1 and also receives personalized advice to consume protein rich foods in close proximity of usual physical activity. All groups receive a standard brochure of the Netherlands or Finnish Nutrition Centre with general information about healthy eating habits. The control group (N=44 at each at each study site) receives no further intervention.

   Main study parameters/endpoints: The primary outcome of this study is change in walk time on the 400 meter walk test. Secondary outcomes are change in dietary intake (including macro- and micronutrients), malnutrition prevalence, physical performance, mobility limitations, muscle strength, body weight and body composition, frailty status, quality of life, and health care costs.

   Statistical analyses:

   The collected data at the two study sites will be pooled together.

   As a result of randomization at study baseline, we assume that groups are equal regarding demographical and socio-economic variables. If this is not the case, we will adjust for differences between groups at baseline. We will adjust for study site (the Netherlands, Finland) and baseline outcome values. We will present unadjusted and adjusted results.

   The main analyses will be based on intention-to-treat principles, but per-protocol analyses will also be conducted as a sensitivity analysis.

   Multiple Imputation (MI) using multivariate Imputation by Chained Equations (MICE) will be used to impute missing cost and effect data. For this, the missing values need to be missing at random.

   The (cost) effectiveness of two intervention groups will be examined against the control group on the primary outcome walk time on the 400 meter walk test. We will compare outcomes between the respective intervention groups and control group separately to determine whether the two interventions are effective (group 1 versus control group; group 2 versus control group).

   We will perform mixed model regression analyses adjusting for confounding variables at baseline and study site as cluster variable. We will not correct for multiple testing but look at the clinical relevance of the outcome.

   In addition, we will perform sensitivity analyses leaving out the participants who took part in the persuasive technology sub-study.

   **** Update June 2020 ****

   Deviation of the protocol

   Due to the worldwide spread of Covid-19, the original protocol of the PROMISS prevention trial has been changed for those participants who were still active in the study during the spread (March 16th - June 1st). In consultation with both Medical Ethical boards from Finland and the Netherlands, and PROMISS' ethical advisor, the following changes were applied:

   March 2020 * Starting from March 16 2020, the final follow-up measurement of 80 participants (out of 276) was postponed until further notice.

   * Participants were informed that they would be invited for the final follow-up measurement when the country-specific governmental regulations allowed it.

   * Participants were requested to stick to their habitual diet (control group) or their intervention diet (both intervention groups).

   April 2020 * Final measurements were resumed (through interview by phone) except for the physical measurements.

   * Dietary intake was assessed in the week prior to the phone call measurement.

   * Self-reported body weight was added to the questionnaire.

   * The physical follow-up measurement was still postponed until further notice.

   May 2020

   * Data collection was continued by means of questionnaires during the phone call measurement in both Finland and the Netherlands.

   June 2020
   * Starting from the beginning of June, the physical measurements at the clinic site were also resumed in both Finland and the Netherlands. Those with no health complaints potentially caused by the coronavirus were allowed to visit the clinic site.
   * The data collection will finish by July 31, 2020.

   We will perform sensitivity analyses excluding those participants who were still active in the study during the spread and thus had their physical follow-up measurement +/- 8 months after the baseline assessment (instead of 6 months).

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 65 years;
* Community-dwelling;
* Lower protein intake defined as both a probability score above a certain cutoff on the protein screener (www.proteinscreener.nl) as well as based on actual protein intake assessed by 24-hour recalls. The protein screener was developed and validated using an extended FFQ among Dutch older adults. The cutoff will be chosen based on results of different studies in which the investigators compare the probability scores of the protein screener with protein intake as measured with food diaries and/or dietary recalls. The investigators will then choose the probability score that is most closely associated with a protein intake < 1.0 g/kg adjusted body weight/day. This probably score reflects older adults with a higher probability on a protein intake < 1.0 g/kg adjusted body weight/d than a general sample of older adults;

Exclusion criteria:

* Inability or unwillingness to provide informed consent
* Not able to eat independently;
* Not able to speak, write and read the Dutch language;
* Current participation to supervised behavioral or lifestyle intervention that intervenes with PROMISS intervention;
* Not able the visit the research site in the following next 6 months;
* Bedridden or wheelchair bound;
* Individuals who do not go outside;
* Diagnosed with severe kidney disease;
* Diagnosed with Parkinson's disease;
* Diagnosed with diabetes mellitus type I;
* Diagnosed with diabetes mellitus type 2 and starting with insulin;
* Current treatment of cancer (with the exception of basal cell carcinoma);
* Vegan diet;
* Severe allergies to certain food products (such as peanuts, gluten);
* Diagnosed with an eating disorder (self-reported);
* Purposefully lost/gained > 3 kg in the past three months
* Heart problems in the past three months (heart attack, angioplasty, heart surgery, stroke or other serious heart disease)
* Not able to complete the 400 meter walk test within 15 minutes (self-reported, and assessed at study baseline).
* Alcohol abuse past 6 months (AUDIT-C ≥ 2);
* Low cognitive status, defined as the mini-mental state examination (MMSE) score ≤ 20
* BMI < 18.5 kg/m2 (self-reported, and assessed at study baseline);
* Overweight, defined as BMI > 32.0 kg/m2 (self-reported, and assessed at study baseline);

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 276 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
6-month change in walk time on a 400 meter walk test | 6 months
  Change in walk time on a 400 meter walk test

SECONDARY OUTCOMES:
6-months change in Physical performance assessed by the Short Physical Performance Battery (SPPB) | 6 months
  SPPB consists of three tests: repeated chair stands test, 4 meter walk test, and tandem stand test. The total score ranges from 0-12. A higher score indicates better physical functioning.
6-month change in hand grip strength | 6 months
  Hand grip strength measured by a hand held dynamometer
6-month change in leg strength | 6 months
  Upper leg strength measured by a measurement chair
6-month change in body composition | 6 months
  Body composition (fat-free mass, skeletal muscle mass and fat mass) will be assessed from bioelectrical impedance using body resistance, reactance, impedance and phase angle. In the Dutch sample only, fat-free mass and fat mass will be directly measured by using densitometry (BODPOD).
3, and 6-moths self-reported mobility limitations (questionnaire) | 3 and 6 months
  Mobility limitations will be assessed by means of a questionnaire; "Because of your health, how much difficulty do you have walking 400 meter?" and "Because of your health, how much difficulty do you have climbing one flight of stairs?" Participants responded using a five level Likert scale: 'No difficulty', 'a little difficulty', 'some difficulty', 'a lot of difficulty', and 'unable to do the activity'.
3, and 6-moths self perceived quality of life | 3 and 6 months
  Quality of life measured using the EuroQol-5D instrument. The EuroQol 5D consists of five questions on a Likert scale (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Answer categories range from (1) 'no problems' to (5) 'unable to'. An additional thermometer for experienced health is scored on a Visual Analogue scale (VAS), ranging from 0-100. The exact point where the line crosses the VAS is the VAS score. The scores are converted to an index value, which facilitates the calculation of quality-adjusted life years (QALYs) that is used to calculate the cost-effectiveness of the study.
Incident frailty assessed by the Fried Frailty Index | 6 months
  Frailty will be determined using the 5 criteria of the Fried Frailty Index:
  * Self-reported unintentional weight loss: >4 kg in past 6 months.
  * Self-reported exhaustion. Based on two self-reported questions from the Center for Epidemiologic Studies Depression scale on exhaustion in the past week at baseline and follow-up: "I felt that everything I did was an effort" and "I could not get going". Scores ranges from 1 'not at all' to 4 'most of the time'. A score of 3 or 4 on either question indicates exhaustion.
  * Weakness: grip strength in the lowest 20% of the study population, adjusted for gender and BMI.
  * Slow walking speed: walk time on the 400 meter walk test in the slowest 20% of the study population, adjusted for gender and height.
  * Low physical activity: Kilocalories expended/wk based on accelerometer data in the lowest quintile of physical activity for each gender.
  Outcome:
  No components:robust
  1 or 2 components:intermediate/prefrail 3 or more components:frail
Incidence of sarcopenia risk | 3 and 6 months
  Incidence of sarcopenia risk will be assessed with the SARC-F questionnaire; how much effort do you experience when 1) lifting and carrying a bag of 4.5 kilo, 2) walking across a room, 3) transferring from a chair or bed, 4) climbing a flight of 10 stairs, and 5) how many times have you fallen in the past year. Answering option include no effort (0 points), a bit of effort (1 point) and a lot of effort (2 points), where a score equal to or greater than 4 is predictive of sarcopenia and poor outcomes.
Incident malnutrition | 6 months
  BMI<22 kg/m2 and unintentional weight loss >5% over 6 months
3, and 6-moths health care costs assessed by questionnaire | 3 and 6 months
  To measure health care costs the investigators will use a modified version of the Resource Utilization in Dementia Questionnaire WIMO. This questionnaire contains questions on hospital admissions, prescribed medicine use, care from health professionals, and use of other health care services in the past three months. These are the domains that the investigators might expect changes in due to the intervention.
3, and 6-month change in body weight | 3 and 6 months
  Body weight (kg) will be measured to the nearest 0,1 kg using a calibrated scale.
Body height | baseline
  Body height (cm) will be measured to the nearest 0.1 cm using a stadiometer.
3, and 6-month change in body mass index (BMI) | 3 and 6 months
  Based on measured weight (measured at baseline and after 6 months) and height (measured at baseline) BMI will be calculated as body weight (kg) divided by height (m) squared.
Dietary intake assesed by three 24-hour recalls | 3 and 6 months
  A 24-hour recall is a structured interview intended to capture detailed information about all foods and beverages consumed by the participant in the past 24 hours. Changes in dietary intake (based on data of the 24-hour recalls) enables to investigate compliance; i.e. higher protein intake indicates higher compliance.
Physical activity | 3 and 6 months
  Physical activity will be objectively assessed by means of an accelerometer (Axivity, AX3) during 7 subsequent days after each clinic visit.

OTHER OUTCOMES:
Effectiveness of persuasive technology sub-study on protein intake | 6 months
  Examine the effect of persuasive technology on adherence to increasing protein intake. A subsample of the Dutch participants will receive a food storage box that can measure which protein rich food products are taken out and a small-size screen (tablet) that provides reminders and nudges. The investigators will test if there are differences in adherence to the interventions between participants who took part in this sub-study and participants who did not.
Microbiota sub-study | 6 months
  The effect of increasing protein intake to at least 1.2 g/kg body weight/d on faecal and oral microbiota composition
Effect of protein intake on satiety and reward responses measured by functional magnetic resonance imaging | 6 months
  To examine the effects of increasing protein intake on food-stimuli related central nervous system satiety and reward responses involved in the regulation of food intake, measured by functional magnetic resonance imaging.
  BOLD fMRI will be used to measure neuronal activity in CNS satiety and reward circuits (including striatum, amygdala, orbitofrontal cortex, insula) in response to visual food stimuli (pictures of food items) and to the actual consumption of food (chocolate milk).

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Visser, Prof., PhD, Study Chair — VU University of Amsterdam
Locations (2):
- University of Helsinki, Helsinki, Finland
- Vrije Universiteit Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Grasso AC, Olthof MR, Reinders I, Wijnhoven HAH, Visser M, Brouwer IA. Effect of personalized dietary advice to increase protein intake on food consumption and the environmental impact of the diet in community-dwelling older adults: results from the PROMISS trial. Eur J Nutr. 2022 Dec;61(8):4015-4026. doi: 10.1007/s00394-022-02896-x. Epub 2022 Jul 5. PMID 35788775
- [Derived] Reinders I, Visser M, Jyvakorpi SK, Niskanen RT, Bosmans JE, Jornada Ben A, Brouwer IA, Kuijper LD, Olthof MR, Pitkala KH, Vijlbrief R, Suominen MH, Wijnhoven HAH. The cost effectiveness of personalized dietary advice to increase protein intake in older adults with lower habitual protein intake: a randomized controlled trial. Eur J Nutr. 2022 Feb;61(1):505-520. doi: 10.1007/s00394-021-02675-0. Epub 2021 Oct 5. PMID 34609621
- [Derived] Reinders I, Wijnhoven HAH, Jyvakorpi SK, Suominen MH, Niskanen R, Bosmans JE, Brouwer IA, Fluitman KS, Klein MCA, Kuijper LD, van der Lubbe LM, Olthof MR, Pitkala KH, Vijlbrief R, Visser M. Effectiveness and cost-effectiveness of personalised dietary advice aiming at increasing protein intake on physical functioning in community-dwelling older adults with lower habitual protein intake: rationale and design of the PROMISS randomised controlled trial. BMJ Open. 2020 Nov 20;10(11):e040637. doi: 10.1136/bmjopen-2020-040637. PMID 33444206